CLINICAL TRIAL: NCT07218354
Title: CSP #2041 - Cessation or Reduction of Alcohol Consumption in VEterans: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of a GLP-1 Receptor Agonist Semaglutide in U.S. Veterans With Alcohol Use Disorder (CRAVE)
Brief Title: Cessation or Reduction of Alcohol Consumption in Veterans: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of a GLP-1 Receptor Agonist Semaglutide in U.S. Veterans With Alcohol Use Disorder
Acronym: CRAVE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2041
Record Dates: First submitted 2025-09-23; First posted 2025-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use Disorder; Semaglutide; Alcohol; GLP-1
MeSH Terms: conditions — Alcoholism | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to either Semaglutide or Placebo injections. The Semaglutide group will be titrated from 0.25 mg up to 2.4 mg/week based on flexible dosing.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants assigned to the placebo group will receive a placebo pen, which mimics the treatment pens by following the same treatment procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Weekly subcutaneous injections of semaglutide up to 2.4 mg/week or maximum tolerated dose. Initial dosing starting at 0.25 for weeks 1-4. Further titration up to 2.4 mg weekly starting at week 5.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Weekly subcutaneous injections of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Weekly subcutaneous injections of semaglutide up to 2.4 mg/week or maximum tolerated dose. Initial dosing starting at 0.25 for weeks 1-4. Further titration up to 2.4 mg weekly starting at week 5.
  Arms: Semaglutide
Drug: Placebo — Weekly subcutaneous injections of placebo.
  Arms: Placebo

SUMMARY:
This clinical trial aims to test the effectiveness and safety of semaglutide, a GLP-1 receptor agonist, in treating moderate to severe alcohol use disorder (AUD) in Veterans. Participants who qualify will be randomly assigned to receive either semaglutide injections or placebo injections over a 28-week period, followed by a 4-week post-treatment safety assessment period. Participants receiving semaglutide will start with a low dose, gradually increasing to a maximum of 2.4 mg per week, depending on their tolerance. The primary measure of success will be a reduction in risky drinking, assessed through a reliable calendar-based interview method called the Timeline Follow-Back (TLFB), a well-validated calendar-based interview technique for recording daily alcohol consumption. The purpose of this research is to gather information on the effectiveness of semaglutide for treating AUD, potentially offering a new and more appealing treatment option.

DETAILED DESCRIPTION:
AUD is one of the leading causes of disability worldwide. The prevalence of AUD is high, affecting 10.9% of US adults and 5.1% of adults worldwide. Oral naltrexone, the most widely prescribed medication for AUD, has a number needed to treat (NNT) to prevent a return to heavy drinking of 12, and thus is only modestly effective. Indeed, less than 2% of adults with AUD receive medication in a given year. Though the Department of Veterans Affairs promotes pharmacotherapy as a best practice, there are over 400,000 Veterans within the Veterans Health Administration (VHA) who have a diagnosis of AUD, with only about 40,000 being actively treated with pharmacotherapy (source: VA Quality Dashboard accessed 1/31/2025). As there have been no new Food and Drug Administration (FDA) approved medications in nearly two decades, there is an urgent need for novel treatments for AUD with superior efficacy and higher patient appeal. Based upon very promising clinical experience, retrospective studies, preclinical data, and recent pilot clinical trial results, the proposed clinical trial is designed to provide definitive evidence regarding the efficacy of the GLP-1 RA, semaglutide, compared to placebo for the treatment of AUD. This research will offer urgently needed information on the efficacy of GLP-1 RAs in the treatment of AUD in a diverse sample and is directly in line with the strategic priorities (SP) for VA Research codified by the Office of Research and Development (ORD) and the National Institute on Alcohol Abuse and Alcoholism (NIAAA).

The proposed study is a randomized, double-blind, placebo-controlled, intent-to-treat, two-arm, parallel, superiority multicenter clinical trial. Veterans with moderate to severe AUD, as diagnosed by DSM-5 criteria, and seeking treatment will be invited to participate. Enrolled participants, meeting eligibility criteria, will be randomized in a 1:1 ratio to receive either semaglutide 2.4 mg or placebo injections using a stratified random block randomization method. The stratification factors are participating site and body mass index (BMI). The study will be conducted in four phases. Phase 1 will be Recruitment, Consent and Screening, Phase 2 will be Randomization and Dose Initiation (the first 4 weeks of treatment), Phase 3 will be the Endpoint Ascertainment Period (24 weeks), and Phase 4 is the Post-Treatment Safety Assessment (4 weeks). Study visits will occur every 4 weeks.

The primary outcome, a reduction in risky drinking, will be assessed by raters at a centralized assessment center (CAC), blinded to treatment assignment, using the Timeline Follow-Back (TLFB). The TLFB is a validated retrospective calendar-based interview technique to record daily alcohol consumption. The TLFB has been widely used in AUD research for its reliability in capturing detailed drinking patterns.

Intervention and Masking Semaglutide 2.4 mg: Participants assigned to the treatment group will undergo 28-week semaglutide treatment. The initial dosing period of 4 weeks (Phase 2) will be used for initiation of 0.25 mg for weeks 1 to 4. Further titration up to 2.4 mg weekly will occur starting at week 5 (Phase 3). Participants should be increased to their maximal tolerable dose. Increases will be considered only after the participant has been on the current dose for 4 weeks. Doses are not to exceed 2.4 mg weekly. Patients may have their dose reduced, maintain their current dose, or have slower titration to ensure tolerability and increase retention in the study. Doses are delivered via a pen, a cartridge-based device that calibrates medication delivery based on the desired dose. An extremely small needle (4-mm, 32-gauge needle - the size of 2 human hairs) is used to deposit the medication subcutaneously.

Placebo: Participants assigned to the placebo group will receive a placebo pen, which mimics the treatment pens under the masking rule by following the same treatment procedure.

Sample Size and Study Duration This study plans to randomize 438 Veterans, with 219 participants assigned to each group. Recruitment is expected to be completed over 32 months.

ELIGIBILITY:
Inclusion Criteria:

* Veteran.
* WHO risk drinking level of Very High or High in the 30 days prior to screening.
* Current diagnosis of moderate or severe AUD (i.e., meeting at least 4 of 11 DSM-5 AUD criteria) based on semi-structured diagnostic exam.
* Able and willing to provide informed consent.

Exclusion Criteria:

Medical and Psychiatric:

* Type 1 diabetes.
* Current serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, borderline or antisocial personality disorder, eating disorder).
* Current DSM-5 diagnosis of a SUD (other than moderate-to-severe alcohol, any nicotine, or mild cannabis use disorders).
* At the time of randomization, moderate-to-severe alcohol withdrawal (Clinical Institute Withdrawal Assessment for Alcohol (CIWA-AR) >8).
* BMI <21 kg/m2.
* Unstable body weight defined as >5% change in body weight (documented or self-report; intentional or not) in the 90 days prior to randomization.
* History of acute or chronic pancreatitis.
* History of diabetic ketoacidosis.
* History of proliferative diabetic retinopathy.
* History of ascites, advanced liver fibrosis, compensated cirrhosis with portal hypertension, decompensated cirrhosis, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or hepatocellular carcinoma (HCC).
* History of stage 3 fibrosis or stage 4 cirrhosis from a liver biopsy.
* Presence of gastroparesis.
* History of acute gallbladder disease in the prior 6 months.
* History of advanced fibrosis or cirrhosis, including (but not limited to) transient elastography (liver stiffness) of >12 kPa, FIB-4 2.67, ELF 9.8, MRE 3.63 kPa.
* History of esophageal varices on endoscopy or imaging.
* History of nodular liver, cirrhosis, splenomegaly, varices or splenic venous shunting or collaterals on prior imaging.
* History or acute alcohol hepatitis (by liver biopsy or elevated bilirubin > 1.5 times the upper limit of normal).
* History of primary biliary cholangitis.
* History of primary sclerosing cholangitis.
* History of autoimmune liver disease.
* History of hemochromatosis.
* History of Wilson's disease.
* History of alpha-10 antitrypsin-related liver disease.
* History of drug-induced liver disease.
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).
* Acute high risk of suicide requiring hospitalization at the time of screening or randomization.
* Medical, psychiatric, behavioral, or logistical conditions which, in the judgment of the Local Site Investigator (LSI) or Sub-Investigator (Sub-I), make it unlikely the participant can participate in or complete the 28-week active phase of the study.
* Recent major cardiovascular event in the 90 days prior to randomization (myocardial infarction, stroke, New York Heart Association class IV heart failure, transient ischemic attack (TIA), or unstable angina.

Laboratory

* Hemoglobin A1c (HbA1c)>10.
* Estimated glomerular filtration rate (eGFR) <30 mL/min.
* Albumin < 3.5 g/dl.
* Aspartate aminotransferase (AST) >3 the Upper Limit of Normal (ULN).
* Alanine aminotransferase (ALT) >3 the ULN.
* Lipase > 2 times the upper limit of normal.
* Alkaline phosphatase > 1.5 times the ULN.
* Total bilirubin > 1.5 times the ULN except with documented Gilbert's syndrome.
* International Normalized Ratio (INR) > 1.3 unless due to anticoagulation therapy.
* Platelet count <150,000/µL unless consistent with baseline and reflects the participant's habitual thrombocyte level, and there was no presence of portal hypertension.
* Hepatitis B surface antigen positive.
* Hepatitis C virus RNA positive - participants treated and cured of hepatitis C must have at least 2 years of negative testing.
* Anti-HIV antibody positive test with uncontrolled or unstable treatment.
* Positive urine drug screen for substances other than cannabis and prescribed medications.
* Positive urine pregnancy test at screening in those considered of childbearing potential.

Concurrent Treatments:

* Current (within the past 30 days) use of pharmacotherapy for AUD (including oral or intramuscular naltrexone, acamprosate, disulfiram, topiramate).
* Known history of prior hypersensitivity reaction to semaglutide, any of the product components, or any other GLP-1 analogue.
* Current (within the past 30 days) use of the following medications with glucose-lowering properties: GLP-1 analogues; sulfonylurea; insulin and insulin products; dipeptidyl peptidase-4 (DPP-4) inhibitors; sodium-glucose cotransporter-2 (SGLT-2) inhibitors or other medications that may interact with semaglutide.
* Recent changes in dose (within 2 months of randomization) of psychiatric medications (i.e., antidepressants, antianxiety, mood stabilizing).

Other

* Pregnant, actively breastfeeding, or female of childbearing potential who is unwilling to use a highly effective method of contraception as defined by the NIH [67].
* Currently enrolled in another therapeutic or investigational clinical trial.
* Participant is incarcerated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-04-28 (Estimated); Study Completion 2029-05-26 (Estimated)

PRIMARY OUTCOMES:
Two-level reduction in the World Health Organization (WHO) risk drinking level | Change from Baseline to Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. The WHO risk drinking levels categorize alcohol consumption into four groups: low (level 1; 0-2.86 standard drinks/day for men; 0-1.43 drinks/day for women), moderate (level 2; 2.87-4.29 standard drinks/day for men; 1.44-2.86 drinks/day for women), high (level 3; 4.3-7.14 standard drinks/day for men; 2.87-4.29 drinks/day for women), and very high (level 4; >7.15 drinks/day for men; >4.3 drinks/day for women). One standard drink is 14g of alcohol. A 2-level reduction, such as moving from very high to moderate risk, is considered a significant clinical improvement.

SECONDARY OUTCOMES:
Adverse events of special interest (Assessing safety and tolerability) | From randomization through week 32.
  Safety and tolerability will be assessed using number of participants (assessing proportion) with adverse events of special interest (AESIs; adverse events reported in >2% of those exposed to the study drug in previous trials).
No heavy drinking days | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment).
Two-level reduction in the World Health Organization (WHO) risk drinking level by Race category | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by race category (White, Black, Other) with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. Each month of the ascertainment phase (weeks 5-28), the WHO risk drinking level will be calculated.
Two-level reduction in the World Health Organization (WHO) risk drinking level by age category (<65, ≥ 65) at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by age category (<65, ≥ 65) at baseline with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. Each month of the ascertainment phase (weeks 5-28), the WHO risk drinking level will be calculated.
Two-level reduction in the World Health Organization (WHO) risk drinking level by psychiatric comorbidity at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with a psychiatric comorbidity at baseline with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. Each month of the ascertainment phase (weeks 5-28), the WHO risk drinking level will be calculated.
Two-level reduction in the World Health Organization (WHO) risk drinking level by presence of other psychiatric treatments (medication and/or psychotherapy) at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with psychiatric treatments (medication and/or psychotherapy) at baseline with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. Each month of the ascertainment phase (weeks 5-28), the WHO risk drinking level will be calculated.
Two-level reduction in the World Health Organization (WHO) risk drinking level by impulsivity category (low, moderate, high) at baseline. | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by impulsivity category (low, moderate, high) at baseline with at least a two-level reduction, from baseline risk level, in WHO risk drinking level. Each month of the ascertainment phase (weeks 5-28), the WHO risk drinking level will be calculated. Impulsivity will be measured by the Barratt Impulsiveness Scale, which is a 30-item self-report instrument designed to access the personality/behavioral construct of impulsiveness. Items are scored on a 4-point scale: Rarely/Never = 1 Occasionally = 2 Often = 3 Almost Always/Always = 4. Total scores range from 30-120, with a higher score indicating a higher level of impulsivity. A score >/= 72 will be classified as high, 52-71 moderate, and < 52 low.
No heavy drinking days by Race category | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by race category (White, Black, Other) with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment).
No heavy drinking days by age category (<65, ≥ 65) at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by age category (<65, ≥ 65) at baseline with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment).
No heavy drinking days by psychiatric comorbidity at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with a psychiatric comorbidity at baseline with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment).
No heavy drinking days by presence of other psychiatric treatments (medication and/or psychotherapy) at baseline | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants with psychiatric treatments (medication and/or psychotherapy) at baseline with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment).
No heavy drinking days by impulsivity category (low, moderate, high) at baseline. | Weeks 5-28. Includes six repeated measurements every 4 weeks from week 5 to 28.
  Number of participants by impulsivity category (low, moderate, high) at baseline with no heavy drinking days. Heavy drinking is defined as >4 standard drinks in a day for men and >3 for women. One standard drink is equal to 14 g of alcohol or approximately 12 oz beer, 5 oz wine, or 1.5 oz of liquor. The data will be derived from the Timeline Follow Back, which is a validated retrospective calendar-based interview technique to record daily alcohol consumption over a specified recall period (since the last assessment). Impulsivity will be measured by the Barratt Impulsiveness Scale, which is a 30-item self-report instrument designed to access the personality/behavioral construct of impulsiveness. Items are scored on a 4-point scale: Rarely/Never = 1 Occasionally = 2 Often = 3 Almost Always/Always = 4. Total scores range from 30-120, with a higher score indicating a higher level of impulsivity. A score >/= 72 will be classified as high, 52-71 moderate, and < 52 low.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Study Chair — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After the main results of this study have been published, de-identified data from the study may be shared with other VA investigators, other Federal health agencies, or academic institutions for the purpose of additional analyses provided this use has been approved by the appropriate VA oversight committee and there is an agreement in place that defines the limits of this use.
  Non-identified study data may be made available to the FDA and Novo Nordisk for medication approval.
Supporting Information: Study Protocol, SAP